CLINICAL TRIAL: NCT05883696
Title: Palliative Care Needs Among Elderly People at Emergency Department
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-05905
Record Dates: First submitted 2023-03-20; First posted 2023-06-01 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Palliative Medicine; Palliative Care; Elderly Person
Keywords: Elderly; palliative care needs; Emergency department; Swedish Palliative Care Guide
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Descriptive patient group: The research nurse will fill in the documents in Swedish Palliative care guide (S-PCG) together with the patient.
  Interventions: Other: Swedish Palliative Care Guide (S-PCG)

INTERVENTIONS:
Other: Swedish Palliative Care Guide (S-PCG) — S-PCG is a care guide that aim to inform best practice and to meet palliative care needs of patients and their families throughout all the time with palliative care needs. The S-PCG support palliative care for adult patients regardless of diagnosis, place of care and if it is early och late palliative care.
  The S-PCG includes three parts
  1. Assessments of palliative care needs
  2. Initiating palliative care 2D. End of life care.
  3. After death. In this study only the first part of the S-PCG will be used.

SUMMARY:
Aim: To assess what proportion of all patients over the age of 75 who seek care at the emergency department have palliative care needs and whether these are documented in the patient's medical record.

Data collection and analysis: Patients over 75 years of age who seek care in an emergency department and are classified as triage 2-4 during initial triage are assessed by a researcher. Patients with dementia or other cognitive dysfunction will be excluded. Two types of data collection are included 1) Swedish Palliative care guide (S-PCG) documents that the researcher fills in together with the patient, 2) data from the patient's medical record, this data is collected according to a special assessment template. Data from the medical record will be collected after the patient left the emergency department.

Data collection is ongoing until 300 patients have been included in the study. Data will be analyzed using descriptive statistics.

Implications: The percentage of previously undetected/documented palliative care needs in emergency departments is relevant for prioritizing general palliative care within e.g. housing for the elderly and primary care S-PCG can be relevant to increase the level of knowledge at these care facilities. If it turns out that many patients have palliative care needs that are not met in the emergency department, health care structures need to ensure that these patients receive help at the right level of care. This would likely mean that the number of emergency visits and hospital admissions (with suffering and reduced quality of life as a result) can be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Classified as triage 2-4

Exclusion Criteria:

* Dementia or other cognitive dysfunction
* Not being able to communicate in Swedish.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients admitted to emergency department in HBG Sweden, aged 75 and above and classified as triage 2-4, without cognitive dysfunction.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Palliative care needs | The study will be ongoing fo up to at year. The S-PCG will be used at 1 time for each included patient.
  The proportion of patients that have palliative care needs that are identified with S-PCG.
Palliative care needs documented in medical records. | The study will be ongoing fo up to at year. The S-PCG will be used at 1 time for each included patient
  The proportion of patients with palliative care need identified with S-PCG as compared to the proportion of palliative care needs documented in the medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Schelin, ass. prof., Principal Investigator — Region Skåne
Locations (1):
- Region Skane, Helsingborg, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No